CLINICAL TRIAL: NCT02949570
Title: Phase 2 Study to Assess Efficacy and Safety of Inecalcitol in Imatinib-Treated Residual Chronic Myeloid Leukaemia: INIM Study
Brief Title: Study to Assess Efficacy and Safety of Inecalcitol in Imatinib-Treated Residual Chronic Myeloid Leukaemia: INIM Study
Acronym: ICT10
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hybrigenics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICT10; 2014-004347-12 (EudraCT Number)
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: CML, Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — inecalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Inecalcitol

INTERVENTIONS:
Drug: Inecalcitol — Prospective open label, non-comparative, multicentre exploratory study. Divided in 2 parts Part1: Inecalcitol treatment will be added to imatinib for 12 months. Part 2: Follow-up after discontinuation of inecalcitol. Imatinib will be maintained for 2 years and then will be stopped for those still in MR4.5. These patients will then be followed for 2 additional years after discontinuation of imatinib.

SUMMARY:
To assess the efficacy of inecalcitol in combination with imatinib in CML patients with molecular residual disease on imatinib monotherapy.

DETAILED DESCRIPTION:
To determine:

* Duration of response
* Progression free survival
* Proportion of responders 2 years after discontinuation of inecalcitol
* Duration of response after discontinuation of inecalcitol and imatinib
* Bone remodelling effect
* Safety of inecalcitol in combination with imatinib
* Quality of Life

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged of at least 18 years at the time of informed consent signature;
* Patients have signed written informed consent;
* ECOG performance status < 2;
* Patients with Philadelphia chromosome positive chronic phase CML and M BCR-ABL transcript positivity (e13a2 or e14a2);
* Treatment with imatinib for more than 2 years (a history of treatment with interferon is tolerated);
* Patient in complete cytogenetic response with BCR-ABL/ABL status between 0.1% International Scale (IS) and 0.01% IS and no BCR-ABL checkpoint in the last six months better than Molecular Response MR4 ( i.e. BCR-ABL ratio < 0.01% IS);
* Women of child bearing potential have a negative pregnancy test prior to first dose and agree to practice effective contraception during the study;
* Fertile men agree to practice effective contraception during the study;
* Patients agree to comply with the study requirements and agree to come to the clinic for required study visits;
* Patients agree to follow medication restrictions during the study;

Exclusion Criteria:

* Expression of unusual BCR-ABL transcripts (other than e13a2 or e14a2);
* Pregnant or lactating women;
* Participating in another clinical trial with any investigative drug within 30 days prior to study enrolment(except for OPTIM imatinib);
* Treatment with interferon within the last 24 months;
* Imatinib dose modification within the last 3 months;
* Prior history of haematopoietic stem cell transplantation;
* Impaired renal function with creatinine clearance < 30 ml/min/1.73m² according to the MDRD formula;
* Hypercalcemia (corrected with albuminemia);
* History of diseases known to be associated with calcium disorders: ongoing hyperparathyroidism, sarcoidosis….;
* Presence or history of symptomatic kidney stones in the last 5 years;
* Current use of drugs known to influence serum calcium (such as thiazide diuretics, teriparatide, calcitonin and multivitamin supplements containing > 400 IU of vitamin D or calcium);
* Current use of digitalis;
* Current use of drugs which could influence bioavailability of inecalcitol (such as magnesium-containing antacids, bile-resin binders);
* Patients with a chronic condition which is not well controlled that, according to the investigator, would interfere with the completion of the study;
* Use of any other experimental drug, therapy or vitamin D supplementation within 30 days of first inecalcitol administration;
* Patients with a mental deficiency preventing proper understanding of trial protocol requirements;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Measure the proportion of responders | 12 months
  Proportion of responder defined as patients achieving MR4.5 (i.e. detectable disease ≤ 0.0032 % BCR-ABLIS or undetectable disease with cDNA with ≥32,000 ABL1 transcripts) at any time within 12 months after the initiation of inecalcitol.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Dufour-Lamartinie, MD, Study Director — Hybrigenics
Locations (1):
- CHU Côte de Nacre, Caen, France

IPD SHARING:
Plan to Share IPD: No